CLINICAL TRIAL: NCT06076161
Title: Effect of Spirulina Platensis Supplementation and Calorie Restriction on Anthropometric, Body Composition, Lipid Profiles, Insulin Resistance, Stress Oxidative Biomarkers In Obese Men: A Randomized Controlled Trial Protocol Study
Brief Title: Spirulina Platensis Supplementation and Calorie Restriction in Obese Men : A Randomized Controlled Trial Protocol Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Adriyan Pramono, Lecturer, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-390
Record Dates: First submitted 2023-09-19; First posted 2023-10-10 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The number of respondents in this study amounted to 32 people. Respondents will be divided into 2 groups, namely the intervention group and the control group. The intervention group will be given spirulina platensis supplements at a dose of 2x2 /hr with a dose per capsule of 450 mg for 4 weeks with education about calorie restriction. The control group will be given placebo 2x2/day for 4 weeks with education on calorie restriction.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will use a randomized controlled trial triple blind study design with a pre-post design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spirulina supplementation and calorie restriction in obese men (Experimental): Respondents will be divided into 2 groups, namely the intervention group and the control group. The intervention group will be given spirulina platensis supplements at a dose of 2x2 /hr with a dose per capsule of 450 mg for 4 weeks with education about calorie restriction.
  Interventions: Dietary Supplement: Spirulina supplementation and calorie restriction in obese men
- Placebo capsules and calorie restriction in obese men (Placebo Comparator): The control group will be given placebo 2x2/day for 4 weeks with education on calorie restriction.
  Interventions: Dietary Supplement: Spirulina supplementation and calorie restriction in obese men

INTERVENTIONS:
Dietary Supplement: Spirulina supplementation and calorie restriction in obese men — The intervention group will be given spirulina platensis supplements at a dose of 2x2 /hr with a dose per capsule of 450 mg for 4 weeks with education about calorie restriction. The control group will be given placebo 2x2/day for 4 weeks with education on calorie restriction.
  Other Names: Placebo capsules

SUMMARY:
The goal of this clinical trial is to evaluate the effects of spirulina platensis supplementation and calorie restriction on anthropometric parameters, body composition, lipid profile, insulin resistance, serum superoxide dismutase (SOD) levels, and serum malondialdehyde (MDA) levels in men with obesity. The main question it aims to answer are:

What is the effect of spirulina platensis supplementation and calorie restriction on anthropometric parameters, body composition, lipid profile, insulin resistance, serum Superoxide Dismutase levels, and serum Malondialdehyde levels in obese individuals?

Participants will be respondents were given spirulina supplements for 30 days with a dose of 2x2 capsules 450mg

Researchers will compare intervention group with placebo group that weren't given spirulina supplementation to see if there is any effects on anthropometric parameters, body composition, lipid profile, insulin resistance, serum Superoxide Dismutase levels, and serum Malondialdehyde levels

DETAILED DESCRIPTION:
Spirulina supplement intervention on subjects with male gender aged 25-55 years, which will be intervened for 4 weeks / 30 days, before the intervention will be taken anthropometric parameters, body composition, lipid profile, insulin resistance, serum Superoxide Dismutase levels, and serum Malondialdehyde levels.

After that, spirulina supplement intervention will be given at a dose of 2x2 / day, and follow-up will be carried out every week, after 30 hours of intervention,spirulina supplement distribution is carried out by research assistants every 2 days.

Will be taken again to conduct anthropometric parameters, body composition, lipid profile, insulin resistance, serum Superoxide Dismutase levels, and serum Malondialdehyde levels.

The aim is to find out if there is an effect of spirulina supplementation on anthropometric parameters, body composition, lipid profile, insulin resistance, serum Superoxide Dismutase levels, and serum Malondialdehyde levels.

ELIGIBILITY:
Inclusion Criteria:

* Male Age 25 - 55 years
* BMI ≥ 30 kg/m2
* Waist Circumference > 90 cm
* Low physical activity (Sedentary life style)
* If taking weight loss supplements are willing to stop the dietary supplements, food or drinks.
* Not undergoing a diet program.

Exclusion Criteria:

* History of kidney disease, atherosclerosis, cancer, and acute infections.
* Post-surgery in the last 3 months.
* Deficit in daily calorie requirement.
* Smoking habit and alcohol dependence.
* Use of hormonal drugs, antidepressant drugs, antibiotics, antidiuretic, glucocorticoids and use of vitamin or mineral supplements in the last three months.
* Refusal to sign the informed consent and in the study if not completing all stages will be excluded.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Obese men
Enrollment: 32 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol | 30 days
  Total Cholesterol in mg/dL
Insulin Resistance - HOMA-IR | 30 days
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) will be measured using fasting blood sugar and blood glucose (both in mg/dL)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 30 days
  Weight in kilograms and height in centimeters. Weight and height will be combined to report BMI in kg/m^2
Serum Superoxide Dismutase (SOD) Levels | 30 days
  SOD levels in U/mL
Serum Malondialdehyde (MDA) Levels | 30 days
  MDA levels in mmol/L
Body Fat Percentage | 30 days
  Body fat percentage in percent

CONTACTS AND LOCATIONS:
Overall Officials: Adriyan Pramono, PhD, Principal Investigator — Department of Nutrition Science, Faculty of Medicine, Diponegoro University, Semarang, Indonesia
Locations (1):
- Central Laboratory, UNDIP Academic Hospital (Rumah Sakit Nasional Diponegoro), Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Based on the consent from the respondent that already written in inform consent, we cannot legally give the information to anyone else

REFERENCES:
- [Background] Fernandez-Sanchez A, Madrigal-Santillan E, Bautista M, Esquivel-Soto J, Morales-Gonzalez A, Esquivel-Chirino C, Durante-Montiel I, Sanchez-Rivera G, Valadez-Vega C, Morales-Gonzalez JA. Inflammation, oxidative stress, and obesity. Int J Mol Sci. 2011;12(5):3117-32. doi: 10.3390/ijms12053117. Epub 2011 May 13. PMID 21686173
- [Background] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Background] Dludla PV, Nkambule BB, Jack B, Mkandla Z, Mutize T, Silvestri S, Orlando P, Tiano L, Louw J, Mazibuko-Mbeje SE. Inflammation and Oxidative Stress in an Obese State and the Protective Effects of Gallic Acid. Nutrients. 2018 Dec 21;11(1):23. doi: 10.3390/nu11010023. PMID 30577684
- [Background] James WP. WHO recognition of the global obesity epidemic. Int J Obes (Lond). 2008 Dec;32 Suppl 7:S120-6. doi: 10.1038/ijo.2008.247. PMID 19136980
- [Background] Chooi YC, Ding C, Magkos F. The epidemiology of obesity. Metabolism. 2019 Mar;92:6-10. doi: 10.1016/j.metabol.2018.09.005. Epub 2018 Sep 22. PMID 30253139
- [Result] Nielsen F, Mikkelsen BB, Nielsen JB, Andersen HR, Grandjean P. Plasma malondialdehyde as biomarker for oxidative stress: reference interval and effects of life-style factors. Clin Chem. 1997 Jul;43(7):1209-14. PMID 9216458
- [Result] Rezaei N, Eftekhari MH, Tanideh N, Mokhtari M, Bagheri Z. Comparison of Antioxidant and Anti-Inflammatory Effects of Honey and Spirulina platensis with Sulfasalazine and Mesalazine on Acetic Acid-Induced Ulcerative Colitis in Rats. Galen Med J. 2019 Jun 10;8:e1095. doi: 10.31661/gmj.v8i0.1095. eCollection 2019. PMID 34466462
- [Result] Zarezadeh M, Faghfouri AH, Radkhah N, Foroumandi E, Khorshidi M, Rasouli A, Zarei M, Mohammadzadeh Honarvar N, Hazhir Karzar N, Ebrahimi Mamaghani M. Spirulina supplementation and anthropometric indices: A systematic review and meta-analysis of controlled clinical trials. Phytother Res. 2021 Feb;35(2):577-586. doi: 10.1002/ptr.6834. Epub 2020 Sep 23. PMID 32967062
- [Result] Naeini F, Zarezadeh M, Mohiti S, Tutunchi H, Ebrahimi Mamaghani M, Ostadrahimi A. Spirulina supplementation as an adjuvant therapy in enhancement of antioxidant capacity: A systematic review and meta-analysis of controlled clinical trials. Int J Clin Pract. 2021 Oct;75(10):e14618. doi: 10.1111/ijcp.14618. Epub 2021 Aug 4. PMID 34235823
- [Result] Moradi S, Ziaei R, Foshati S, Mohammadi H, Nachvak SM, Rouhani MH. Effects of Spirulina supplementation on obesity: A systematic review and meta-analysis of randomized clinical trials. Complement Ther Med. 2019 Dec;47:102211. doi: 10.1016/j.ctim.2019.102211. Epub 2019 Oct 17. PMID 31780031
- [Result] Hernandez-Lepe MA, Lopez-Diaz JA, Juarez-Oropeza MA, Hernandez-Torres RP, Wall-Medrano A, Ramos-Jimenez A. Effect of Arthrospira (Spirulina) maxima Supplementation and a Systematic Physical Exercise Program on the Body Composition and Cardiorespiratory Fitness of Overweight or Obese Subjects: A Double-Blind, Randomized, and Crossover Controlled Trial. Mar Drugs. 2018 Oct 1;16(10):364. doi: 10.3390/md16100364. PMID 30275428
- [Result] DiNicolantonio JJ, Bhat AG, OKeefe J. Effects of spirulina on weight loss and blood lipids: a review. Open Heart. 2020 Mar 8;7(1):e001003. doi: 10.1136/openhrt-2018-001003. eCollection 2020. PMID 32201580
- See also: Inflammation, oxidative stress, and obesity — https://pubmed.ncbi.nlm.nih.gov/21686173/
- See also: Obesity: global epidemiology and pathogenesis — https://pubmed.ncbi.nlm.nih.gov/30814686/
- See also: Inflammation and Oxidative Stress in an Obese State and the Protective Effects of Gallic Acid — https://pubmed.ncbi.nlm.nih.gov/30577684/
- See also: The epidemiology of obesity — https://pubmed.ncbi.nlm.nih.gov/30253139/
- See also: Comparison of Antioxidant and Anti-Inflammatory Effects of Honey and Spirulina platensis with Sulfasalazine and Mesalazine on Acetic Acid-Induced Ulcerative Colitis in Rats — https://pubmed.ncbi.nlm.nih.gov/34466462/
- See also: Anti-inflammatory and antithrombotic properties of polar lipid extracts, rich in unsaturated fatty acids, from the Irish marine cyanobacterium Spirulina subsalsa — https://doi.org/10.1016/j.jff.2022.105124
- See also: Impact of spirulina supplementation on obesity-related metabolic disorders: A systematic review and meta-analysis of randomized controlled trials — https://cris.usil.edu.pe/en/publications/impact-of-spirulina-supplementation-on-obesity-related-metabolic-